CLINICAL TRIAL: NCT00927771
Title: Efficacy & Safety of Azelaic Acid 15% Gel vs. Hydroquinone 4% Cream in the Treatment of Melasma
Brief Title: Azelaic Acid Versus Hydroquinone in Melasma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Callender Center for Clinical Research (Other)
Responsible Party: Valerie D. Callender, MD, Callender Center for Clinical Research
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 09-01-01
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Melanosis
Keywords: melanosis; melasma; azelaic acid; hydroquinone
MeSH Terms: conditions — Melanosis | interventions — Hydroquinones; hydroquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azelaic Acid (Experimental)
  Interventions: Drug: azelaic acid gel
- Hydroquinone (Active Comparator)
  Interventions: Drug: hydroquinone cream

INTERVENTIONS:
Drug: azelaic acid gel — azelaic acid 15% gel twice a day for 6 months
  Other Names: Finacea Gel
  Arms: Azelaic Acid
Drug: hydroquinone cream — hydroquinone 4% cream twice a day for 6 months
  Other Names: Claripel; Lustra
  Arms: Hydroquinone

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of Azelaic Acid Gel to Hydroquinone Cream in the treatment of melasma.

DETAILED DESCRIPTION:
Melasma is a chronic condition in which dark areas appear on the forehead, cheeks, and upper lips. Hydroquinone is a skin lightener (or fade cream) and is one of the most commonly used medications for the treatment of melasma. Azelaic acid gel is currently used to treat acne and rosacea.

ELIGIBILITY:
Inclusion Criteria:

* must have stable moderate-severe epidermal or mixed melasma involving the face
* all races
* males and females
* persons taking birth control medication, hormone replacement therapy or any other hormone altering medication may participate only if they have not started or stopped the medication within the last 3 months

Exclusion Criteria:

* if the person has only dermal melasma
* pregnancy, breastfeeding, a positive pregnancy test in the office or plans to become pregnant
* a known allergy or sensitivity ot azelaic acid or hydroquinone
* the use of photosensitizing medications (ex. tetracycline) within 3 months of the study.
* starting or stopping hormonal medication within 3 months
* chemical peels, microdermabrasion, or laser treatment within 6 months
* worsening or improving melasma

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of melasma | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Valerie D Callender, MD, Principal Investigator — Howard University
Locations (1):
- Callender Center for Clinical Research, Mitchellville, Maryland, United States